CLINICAL TRIAL: NCT02207205
Title: A Study to Determine Variability in the Measurement of Whole Blood Clotting Time (WBCT) Between Blood Drawn From Indwelling Catheters and Direct Venipuncture
Brief Title: Variability in the Measurement of WBCT Between Blood Drawn From Indwelling Catheters and Direct Venipuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Perosphere Pharmaceuticals Inc, a wholly owned subsidiary of AMAG Pharmaceuticals, Inc. (Industry)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PER977-01-006
Record Dates: First submitted 2014-07-28; First posted 2014-08-04 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Catheter vs venipuncture blood samples (Other): Evaluation of whether there is any difference in results of whole blood clotting time in blood samples drawn from an indwelling catheter versus direct venipuncture
  Interventions: Drug: Blood drawn from indwelling catheters versus direct venipuncture

INTERVENTIONS:
Drug: Blood drawn from indwelling catheters versus direct venipuncture — Evaluation of the source of blood samples on whole blood clotting time

SUMMARY:
1. Determine if there is any difference between the whole blood clotting time results obtained from blood drawn from indwelling catheters and direct venipuncture
2. Determine the intra-subject variability in both procedures

DETAILED DESCRIPTION:
No investigational products were administered to any subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated, written informed consent (Institutional Review Board [IRB]-approved informed consent form [ICF]).
2. Healthy (as determined by medical history) male and female subjects aged 18 to 65 years (inclusive) with suitable veins for venipuncture.

Exclusion Criteria:

1. Healthy subjects who do not conform to the above inclusion criteria.
2. Healthy subjects who cannot communicate reliably with the Investigator.
3. History of major bleeding or major trauma within the past 6 months
4. Healthy volunteer with a propensity to bleed (i.e. due to recent trauma, recent surgery, peptic ulcer, active or recent gastrointestinal bleeding or bleeding from hemorrhoids).
5. Significant infection or known inflammatory process within 2 weeks of screening.
6. Treatment with any investigational products or therapies within 30 days (or 5 half lives, whichever is greater) prior to screening.
7. Received non-steroidal anti-inflammatory drug (NSAID) or medications (including aspirin) with a direct effect on hemostasis within 7 days of testing
8. Unwillingness or inability to comply with procedures required in this protocol.
9. Subjects who are concurrently enrolled in any other clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Whole blood clotting time results from blood drawn from indwelling catheters and direct venipuncture | single day sampling
  Comparison of results in whole blood clotting time from blood sampled by direct venipuncture and from indwelling catheters as assessed by multiple technicians

CONTACTS AND LOCATIONS:
Overall Officials: Robert Noveck, MD, Principal Investigator — Duke Clinical Research Unit
Locations (1):
- Duke Clinical Research Unit, Durham, North Carolina, United States